CLINICAL TRIAL: NCT04377295
Title: Study of Retinal and Vascular Features by Optical Coherence Tomography and Optical Coherence Tomography Angiography After Intravitreal Injections of Ranibizumab in Radiation Maculopathy
Brief Title: Evaluation of Retinal and Vascular Features in Radiation Maculopathy After Intravitreal Injections of Ranibizumab
Status: Completed | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Gilda Cennamo, Principal Investigator, Federico II University
Other Study IDs: PT1034/20
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Radiation Maculopathy
MeSH Terms: interventions — Ranibizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Ranibizumab 0.5Mg/0.05Ml Oph Inj — All patients received one monthly intravitreal injection of Ranibizumab (0.5 mg/0.05 ml) through the pars plana under aseptic conditions until maximum visual acuity was achieved and there was no sign of macular edema at optical coherence tomography

SUMMARY:
This study evaluates the retinal and vascular features in patients with radiation maculopathy under the effects of Ranibizumab intravitreal injections using optical coherence tomography and optical coherence tomography angiography.

DETAILED DESCRIPTION:
The radiation maculopathy is a consequence of radiotherapy for treatment of choroidal melanoma. The radiation maculopathy is characterized by the compromission of the macular microvasculature that can lead to the leakage, lipid exudates, hemorrhages, teleangiectasie, macular edema, non perfusion areas with consequent significant impaiment of visual acuity.

Ranibizumab is a vascular endothelial growth factor antagonist and it represents an efficacy treatment acting on vascular hyperpermeability. The optical coherence tomography and optical coherence tomography angiography represent novel and non-invasive diagnostic techniques that allow a detailed analysis of retinal and vascular features. The study evaluates the changes in optical coherence tomography and optical coherence tomography angiography parameters at baseline and after intravitreal injections of Ranibizumab at the last follow up to one year in patients affected by radiation maculopathy.

ELIGIBILITY:
Inclusion Criteria:

* age older than 40 years
* diagnosis of radiation maculopathy
* treatment-naïve with Ranibizumab
* absence of other vitreoretinal and vascular retinal diseases

Exclusion Criteria:

* age younger than 40 years
* No diagnosis of radiation maculopathy
* previous treatments with Ranibizumab
* presence of vitreoretinal and vascular retinal diseases

Ages: 40 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: The participans were older than 40 years with diagnosis of radiation maculopathy. They did not present other ophthalmological diseases.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2012-10-30 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Study of retinal and vascular features in pazients affected by radiation maculopathy after intravitreal injections of Ranibizumab | one year
  The effectiveness of Ranibizumab injections for treating radiation maculopathy using optical coherence tomography (OCT).
  The parameter analyzed by OCT was: Central Macular Thickness (micron).
Study of retinal and vascular features in patients affected by radiation maculopathy after intravitreal injections of Ranibizumab | one year
  The effectiveness of Ranibizumab injections for treating radiation maculopathy using optical coherence tomography angiography (OCTA).
  The parameter analyzed by OCTA was: retinal vessel density (%)

CONTACTS AND LOCATIONS:
Overall Officials: Gilda Cennamo, Principal Investigator — Federico II University